CLINICAL TRIAL: NCT06143254
Title: The Effect of Using Symbolic Gestures on the Speech and Language Development in Prelinguistic Children Born With Cleft Palate
Brief Title: Effect of Infant Sign Training on Speech-language Development
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2022-0581
Record Dates: First submitted 2023-11-10; First posted 2023-11-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cleft Palate Children
Keywords: cleft palate; gesture; speech and language development; therapy
MeSH Terms: conditions — Cleft Palate; Gestures; Speech

STUDY DESIGN:
Intervention Model Description: The trial is a two-centre, randomized, parallel-group, longitudinal, controlled trial. Treatment allocation is in a 1:1:1:ratio. Children are randomized to either an infant sign training group (IST group), a verbal training group (VT group) or no intervention control group (C group). The aim is to demonstrate superiority of the active intervention (IST group) compared with control (VT group and C group).
Who Masked: Investigator, Outcomes Assessor
Masking Description: All tests and recordings will be performed by two SLPs of the research group with experience in the diagnosis and treatment of speech and language disorders in children with CP±L. The annotation, analysis and scoring will be performed by the same SLPs. Both raters will analyze 100% of the video-recordings to calculate inter-rater reliability. To calculate intra-rater reliability, both raters will re-assess 20% of the recordings. The raters will not provide intervention to any of the included children and caregivers. They will be blinded for group allocation of the child and caregivers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Symbolic Gesture Training Group (Experimental): Caregivers of children who are assigned to the SGT group will participate in three caregiver training meetings to learn how to use infant signing in combination with verbal training to promote the speech and language development of their child. These meetings will take place 1 month (meeting 1), 2 months (meeting 2) and 3 months (meeting 3) after baseline assessments are performed (T0). Each meeting will take two hours. After the first training session (meeting 1), caregivers will start using the symbolic gestures to support verbal in- and output at home with their child.
  Interventions: Behavioral: Infant sign training
- Verbal Training Group (Active Comparator): Caregivers of children who are assigned to the VT group will participate in three caregiver training meetings to learn how to use verbal training to promote the speech and language development of their child. These meetings will take place 1 month (meeting 1), 2 months (meeting 2) and 3 months (meeting 3) after baseline assessments are performed (T0). Each meeting will take two hours. After the first training session (meeting 1), caregivers will start using supporting verbal in- and output at home with their child.
  Interventions: Behavioral: Verbal training
- No Intervention Control Group (No Intervention): Standard clinical care at this moment at the Cleft Palate Teams of the University Hospitals of Ghent and Leuven includes providing information to caregivers about speech-language development and encouraging caregivers to communicate with their children. This information will be orally provided by an SLP during a standard clinical appointment at the cleft team at the age of 12 months. A brochure including this information will be provided. Caregivers of children who will be assigned to group C will have the opportunity to receive the most effective intervention (SGT or VT) after finishing the study.

INTERVENTIONS:
Behavioral: Infant sign training — Training session 1: Information is given about what infant signs are, how they originated, how speech and (gestural) language develop in young children with CP ± L, the possible advantages of using infant signs and tips for success. Twelve signs are chosen to start with: six narrative signs (mostly object concepts) and six steering signs (mostly non-object concepts). Training session 2: Experiences with using infant signs at home are shared, repetition of the 12 infant signs and tips for success are discussed. Another 12 signs are chosen to add to the repertoire the caregivers can use, based on caregiver input. Training session 3: The same as training session 2. The content is based on the input the caregivers experience. Another 12 signs are chosen to add to the repertoire the caregivers can use, based on caregiver input. Reading aloud while using infant signs is shown and practiced.
  Arms: Symbolic Gesture Training Group
Behavioral: Verbal training — Training session 1: Information is given about how speech and language develop in young children with CP ± L and how caregivers can support their child during this development Tips for success and suggestions on how to use these supportive verbal techniques at home are discussed. Training session 2: Experiences with using supportive verbal techniques at home are shared and supportive verbal techniques repeated. Information is provided about how children learn new words and tips for success are expanded. Training session 3: The same as training session 2. The content is based on the input the caregivers experience. Additionally, advances of reading aloud are discussed and reading aloud is practiced.
  Arms: Verbal Training Group

SUMMARY:
Children born with a cleft lip and palate (CLP) are known to be at risk for speech-language disorders that impact academic and social emotional growth. Even at very young ages (<3 years), speech-language disorders are already observed. It is hypothesized that speech-language intervention delivered before the age of 3 years old could decrease the impact of CLP on speech-language development. This would result in a decreased need for speech-language therapy on the long-term and a reduced burden of care on children, families and health services. However, no evidence is yet available to support any specific model of early speech-language intervention in this population. Consequently, no standardized clinical practice guidelines are available yet. Symbolic gesture training in combination with verbal input expands the natural communication of young children including multimodal speech-language input (i.e., verbal and manual input) via caregivers who act as co-therapists. To contribute to the evidence-based practice in the field of cleft speech therapy, this research project aims to determine the effectiveness and feasibility of symbolic gesture training in one-year old children with CLP by comparing different intervention approaches based on perceptual, psychosocial and qualitative outcome measures.

DETAILED DESCRIPTION:
Children with CP±L are known to be at risk for speech-language delays that impact educational and social-emotional growth. Early intervention in this population mostly focuses on improving verbal input via caregivers or professionals without including a multimodal language input. As stated above, no evidence is yet available for the effectiveness and feasibility of early intervention based on symbolic gesture training in combination with verbal input to improve speech-language skills in young children with CP±L. To contribute to the evidence-based practice in the field of early cleft palate speech intervention, this research project will focus on the effectiveness of symbolic gesture training in one-year old children with CP±L by comparing different intervention approaches based on quantitative and qualitative outcome measures. This project meets the need to evaluate the impact of early intervention on speech-language outcomes in children with CP±L as proposed by several researchers based on reviews regarding this topic.

The primary objective is to explore if children with CP±L who are enrolled in symbolic gesture training to support verbal in- and output at the age of 12 months have increased receptive and expressive language skills compared to children with CP±L who are enrolled in verbal training or not involved in any intervention at all.

The secondary objectives are:

2.1 To explore if children with CP±L who are enrolled in symbolic gesture training at the age of 12 months have improved speech skills, compared to children with CP±L who are enrolled in verbal training or not involved in any intervention at all; 2.2 To explore if children with CP±L who are enrolled in symbolic gesture training at the age of 12 months demonstrate more gesture use, compared to children with CP±L who are enrolled in verbal training or not involved in any intervention at all; 2.3 To explore if caregivers of children with CP±L who are enrolled in symbolic gesture training when their child is 12 months of age provide more frequent and more complex linguistic input to their child's utterances compared to caregivers of children with CP±L who are enrolled in verbal training or not involved in any intervention at all.

ELIGIBILITY:
Inclusion Criteria:

* Born with cleft palate (with or without cleft lip)
* Having Dutch as mother tongue

Exclusion Criteria:

* syndromic cleft
* more than mild hearing loss (i.e. > 40dB hearing threshold bilaterally)
* neurosensory hearing loss
* cognitive delay
* motor delay

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Receptive language level based on language test | 12 months
  To verify the receptive language level, the Dutch Nonspeech Test will be used at T0 and T1. This standardized test observes, scores and judges communication conditions and first verbal and non-verbal communication in the age range of 12 to 21 months. At T2, the Schlichting Test of Language Comprehension and Language Production will be used. This standardized test measures receptive and expressive language development starting from 24 months of age.
  This outcome measure will be expressed in percentiles.
Expressive language level based on language test | 12 months
  To verify the expressive language level, the Dutch Nonspeech Test will be used at T0 and T1. This standardized test observes, scores and judges communication conditions and first verbal and non-verbal communication in the age range of 12 to 21 months. At T2, the Schlichting Test of Language Comprehension and Language Production will be used. This standardized test measures receptive and expressive language development starting from 24 months of age.
  This outcome measure will be expressed in percentiles.
Total language level based on caregiver report | 12 months
  Caregivers will complete the Dutch version of the MacArthur Communicative Development Inventory, 'words and signs' (T0 and T1) or 'words and sentences' (T2). These standardized questionnaires evaluate word comprehension and production, the use of signs by the child, and grammatical development.
  This outcome measure will be expressed in percentiles.

SECONDARY OUTCOMES:
Communicative acts produced by the child | 12 months
  The communicative acts of the child will be analyzed based on a video recording of 30 minutes free play with four standardized toy sets (i.e., a farm, a house, cutlery, and vehicles) between the child and caregiver at T0, T1 and T2. Each potential communicative act of the child will be annotated by the means of communication (eye contact, gesture or vocalization; vocalization will be identified as non-canonical, canonical or word).
  This outcome measure will be expressed in the total number of communicative acts produced by the child.
Communicative acts produced by the caregiver | 12 months
  The communicative acts of the caregiver will be analyzed based on a video recording of 30 minutes free play with four standardized toy sets (i.e., a farm, a house, cutlery, and vehicles) between the child and caregiver at T0, T1 and T2. Each potential communicative act of the caregiver will be annotated by the means of communication (eye contact, gesture or vocalization).
  This outcome measure will be expressed in the total number of communicative acts produced by the caregiver.
Articulatory precision of the child | 12 moths
  Based on the vocalizations of the child, the Percentage Consonants Correct will be determined. This outcome measure is expressed in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Kristiane Van Lierde, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No
Data are stored in REDCap, an electronic data capture system (Harris et al., 2019). The research is carried out in accordance with the information security policy of Ghent University. Personal data are pseudo-anonymized at the level of data collection and anonymized at the level of data analysis. A separate file is created with the key to the code assigned to each participant. This file is stored separately from the other databases and is only accessible to the first and last authors or to the appointed replacement. Only anonymized data are used for analysis and in any type of documentation, reports or publications concerning this study.

REFERENCES:
- [Background] De Ryck M, Van Lierde K, Alighieri C, Hens G, Bettens K. A protocol for a randomized-controlled trial to investigate the effect of infant sign training on the speech-language development in young children born with cleft palate. Int J Lang Commun Disord. 2023 Nov-Dec;58(6):2212-2221. doi: 10.1111/1460-6984.12920. Epub 2023 Jun 28. PMID 37376898
- [Background] Lancaster HS, Lien KM, Chow JC, Frey JR, Scherer NJ, Kaiser AP. Early Speech and Language Development in Children With Nonsyndromic Cleft Lip and/or Palate: A Meta-Analysis. J Speech Lang Hear Res. 2019 Dec 13;63(1):14-31. doi: 10.1044/2019_JSLHR-19-00162. Print 2020 Jan 22. PMID 31841365
- [Background] Scherer NJ, Boyce S, Martin G. Pre-linguistic children with cleft palate: growth of gesture, vocalization, and word use. Int J Speech Lang Pathol. 2013 Dec;15(6):586-92. doi: 10.3109/17549507.2013.794475. Epub 2013 Sep 27. PMID 24073662
- [Background] Lane H, Harding S, Wren Y. A systematic review of early speech interventions for children with cleft palate. Int J Lang Commun Disord. 2022 Jan;57(1):226-245. doi: 10.1111/1460-6984.12683. Epub 2021 Nov 12. PMID 34767284
- [Background] Bessell A, Sell D, Whiting P, Roulstone S, Albery L, Persson M, Verhoeven A, Burke M, Ness AR. Speech and language therapy interventions for children with cleft palate: a systematic review. Cleft Palate Craniofac J. 2013 Jan;50(1):e1-e17. doi: 10.1597/11-202. Epub 2012 Mar 20. PMID 22433039
- [Background] Chapman KL, Hardin-Jones M, Halter KA. The relationship between early speech and later speech and language performance for children with cleft lip and palate. Clin Linguist Phon. 2003 Apr-May;17(3):173-97. doi: 10.1080/0269920021000047864. PMID 12858838
- [Background] Frey JR, Kaiser AP, Scherer NJ. The Influences of Child Intelligibility and Rate on Caregiver Responses to Toddlers With and Without Cleft Palate. Cleft Palate Craniofac J. 2018 Feb;55(2):276-286. doi: 10.1177/1055665617727000. Epub 2017 Dec 14. PMID 29351026